CLINICAL TRIAL: NCT03098420
Title: Dose Escalation of Dexamethasone to Increase Duration of Transversus Abdominal Plane Block Following Cesarean Section: A Prospective Randomized Double-Blinded Clinical Study
Brief Title: Dose Escalation of Dexamethasone to Increase Duration of Transversus Abdominal Plane Block Following Cesarean Section
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low enrollment; recruitment challenges due to competing studies in women and infant center
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Joel Feinstein, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F160421006
Record Dates: First submitted 2017-03-13; First posted 2017-03-31 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Post Surgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Calcium Dobesilate; Ropivacaine; Morphine; Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to 1 of 3 groups. They will be assigned to a group prior to being brought back to the operating room. The anesthesia team in the OR will take an envelope that has which group the patient will be randomly assigned to and they will perform the TAP block with the respective dose of dexamethasone. The anesthesia team that performs the block, along with the supervising PI or sub-investigator, will be blinded to the medication in the injectate
Who Masked: Participant, Investigator
Masking Description: The anesthesia team that performs the block, along with the supervising PI or sub-investigator, will be blinded to the medication in the injectate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Placebo Comparator): 20 patients. Each patient will receive postoperative bilateral TAP blocks (20mL of ropivacaine) and 1mL of normal saline bilaterally (control) with standard intrathecal bupivacaine and morphine.
  Interventions: Drug: Ropivacaine (TAP blocks); Drug: Morphine; Drug: Bupivacaine Hydrochloride; Drug: Normal saline 1ml
- 2mg Dexamethasone (Active Comparator): 20 patients. Each patient will receive postoperative bilateral TAP blocks (20mL of 0.5% ropivacaine) with 0.5 mL (2mg) of dexamethasone and 0.5 ml of normal saline split between 2 sides with standard intrathecal bupivacaine and morphine.
  Interventions: Drug: 2mg Dexamethasone; Drug: Ropivacaine (TAP blocks); Drug: Morphine; Drug: Bupivacaine Hydrochloride; Drug: Normal saline 0.5ml
- 4mg Dexamethasone (Active Comparator): 20 patients. Each patient will receive postoperative bilateral TAP blocks (20mL of 0.5% ropivacaine) with 20mL of 0.5% ropivacaine) and 1 mL (4mg) of dexamethasone between 2 sides with standard intrathecal bupivacaine and morphine.
  Interventions: Drug: 4mg Dexamethasone; Drug: Ropivacaine (TAP blocks); Drug: Morphine; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: 2mg Dexamethasone — 0.5 mL (2mg) of dexamethasone and 0.5 ml of normal saline
  Other Names: Baycadron, Maxidex, Decadron
  Arms: 2mg Dexamethasone
Drug: 4mg Dexamethasone — 1 mL (4mg) of dexamethasone
  Other Names: Baycadron, Maxidex, Decadron
  Arms: 4mg Dexamethasone
Drug: Ropivacaine (TAP blocks) — 20mL of 0% ropivacaine with 20mL of 0.5% ropivacaine
Drug: Morphine
Drug: Bupivacaine Hydrochloride
Drug: Normal saline 1ml — 1.0 ml of normal saline split between 2 sites with standard intrathecal bupivacaine and morphine
  Arms: Control Group
Drug: Normal saline 0.5ml — 0.5 ml of normal saline split between 2 sites with standard intrathecal bupivacaine and morphine
  Arms: 2mg Dexamethasone

SUMMARY:
The study aims to improve the care of the obstetric population after cesarean section and improve total patient satisfaction by improving post-surgical pain control with the use of dexamethasone in combination with bilateral TAP blocks. The investigators will utilize a dose-escalation of dexamethasone in the TAP block to observe its effects at specific small doses. It is the hope of the investigator that the studied technique would become utilized routinely for the obstetric population following cesarean section.

The investigators hope to show that the addition of dexamethasone in bilateral TAP blocks will prolong the duration of the block in a dose-dependent fashion. The investigators hope to improve post-operative pain following cesarean section, increase duration of TAP block with use of dexamethasone, decrease overall pain scores in the first 24-48 hours, and decrease opioid requirements after cesarean section.

The primary endpoint will be estimation of duration of TAP block, being assessed within 48 hours after surgery. Secondary endpoints will include pain scores both in PACU and on the floor, average pain scores, time until first opioid administration, total opioid consumption in first 48 hours, use of PONV medications, and overall patient satisfaction.

DETAILED DESCRIPTION:
Preoperatively: informed consent will be obtained by a member of this study. The patients will be screened for inclusion/exclusion criteria on day of procedure, and then the participants will be randomized to one of three groups.

Intraoperatively: The anesthesia team involved with care of patient in the operating room will provide routine anesthesia care during the cesarean section including neuraxial anesthesia with intrathecal bupivacaine and morphine.

After completion of the procedure, the patients will receive bilateral TAP block procedure while still in OR. All blocks will include 20mL of 0.5% ropivacaine, and the patients will be randomly assigned a specific dose of dexamethasone at 0mg (given normal saline as control), 2mg, or 4mg. The resident or attending physician supervising the block will be investigators of the study, and they along with the residents performing the blocks will be blinded to the amount of dexamethasone in the injectate.

Postoperatively: The patients will then be monitored in the PACU for approximately 30-60 minutes and then subsequently monitored on an inpatient floor. Pain scores, time until first opioid dose, total opioid requirement will be assessed and recorded. In PACU, these will be recorded every 15-30 minutes. On the inpatient floor, these will be recorded every 6 hours.

Pain scores, average pain scores in first 48 hours, total opioid consumption, time until first opioid use, and PONV medication requirement will also be recorded. These will be recorded by review of the electronic medical record.

Satisfaction scores and estimation of TAP block duration will be assessed and recorded by anesthesia personnel approximately 48 hours post-operatively; these will be subjective evaluations recorded between 24-38 hours postoperatively. The patients will be asked to estimate how long they felt the block lasted. For satisfaction scores, patients will rate their satisfaction subjectively on a scale of 1-10.

Statistical Analysis: all demographic and clinical variables with continuous measures will be expressed as means and standard deviations; categorical factors will be expressed as proportions. For non-normal data, the medians and inter quartile ranges will be displayed. The distribution of the continuous factors will be examined using the Kolmogorov-Smirnov test. For data that are normally distributed, one-way ANOVA will be used to compare groups of data. For data that are not normally distributed, the Kruskal-Wallis test will be used for comparisons. Chi-square and Fisher's exact tests will be used to analyze categorical data. For all comparisons, a value of p < 0.05 will be considered statistically significant.

Statistical analyses will be performed using SAS for Windows, version 9.2. One-way ANOVA (or the Kruskal-Wallis test, as appropriate) will be used to compare duration of TAP block for the three groups. Linear regression will also be used to test the relationship between duration of block and dexamethasone dose, while controlling for relevant clinical and demographic variables.

One-way ANOVA (or the Kruskal-Wallis test) will be used to compare the groups on post-operative pain scores, opioid requirements, and patient satisfaction scores.

Statistical Power and Sample Size Estimates: Approximately 69 subjects (23 per group) are expected to be enrolled in this study. Given this sample size and assuming that the average duration of TAP block is 18 hours for the control group, 22 hours for the 2 mg of dexamethasone group, and 24 hours for the 4 mg of dexamethasone group, this study will have approximately 80.9% power to detect a difference in block duration, assuming a common standard deviation of 6 hours. If the variability in block time is smaller than 6 hours, this study will have greater power.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing cesarean section delivery.
2. Patients classified as American Society of Anesthesiology (ASA) class II or III.

   1. ASA II: mild systemic disease, pregnancy
   2. ASA III: severe systemic disease
3. Women ≥ 18 years old
4. Neuraxial anesthesia (spinal) to be used as anesthetic technique intraoperatively for cesarean section (this is the UAB Anesthesiology standard of care).

Exclusion Criteria:

1. Any patient not classified as an ASA I or II.
2. General Anesthesia or neuraxial anesthesia with epidural used as anesthetic techniques for cesarean section.
3. Allergy/intolerance to local anesthetic or steroids.
4. Pre-existing neurological and/or anatomical deficit that would preclude regional block.
5. Coexisting coagulopathy such as hemophilia or von Willebrand Disease
6. BMI > 40.
7. Emergency Cesarean Sections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females undergoing cesarean section delivery
Enrollment: 29 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Feinstein, MD, Principal Investigator — Anesthesiology ad Perioperative Medicine
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: 20 patients. Each patient will receive postoperative bilateral TAP blocks (20mL of ropivacaine) and 1mL of normal saline bilaterally (control) with standard intrathecal bupivacaine and morphine.
  Ropivacaine (TAP blocks): 20mL of 0% ropivacaine with 20mL of 0.5% ropivacaine
  Morphine
  Bupivacaine Hydrochloride
  Normal saline 1ml: 1.0 ml of normal saline split between 2 sites with standard intrathecal bupivacaine and morphine
- 2mg Dexamethasone: 20 patients. Each patient will receive postoperative bilateral TAP blocks (20mL of 0.5% ropivacaine) with 0.5 mL (2mg) of dexamethasone and 0.5 ml of normal saline split between 2 sides with standard intrathecal bupivacaine and morphine.
  2mg Dexamethasone: 0.5 mL (2mg) of dexamethasone and 0.5 ml of normal saline
  Ropivacaine (TAP blocks): 20mL of 0% ropivacaine with 20mL of 0.5% ropivacaine
  Morphine
  Bupivacaine Hydrochloride
  Normal saline 0.5ml: 0.5 ml of normal saline split between 2 sites with standard intrathecal bupivacaine and morphine
- 4mg Dexamethasone: 20 patients. Each patient will receive postoperative bilateral TAP blocks (20mL of 0.5% ropivacaine) with 20mL of 0.5% ropivacaine) and 1 mL (4mg) of dexamethasone between 2 sides with standard intrathecal bupivacaine and morphine.
  4mg Dexamethasone: 1 mL (4mg) of dexamethasone
  Ropivacaine (TAP blocks): 20mL of 0% ropivacaine with 20mL of 0.5% ropivacaine
  Morphine
  Bupivacaine Hydrochloride
Period: Overall Study
Arm/Group | Control Group | 2mg Dexamethasone | 4mg Dexamethasone
Started | 7 | 9 | 13
Completed | 7 | 9 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | 2mg Dexamethasone | 4mg Dexamethasone | Total
Number analyzed (Participants) | 7 | 9 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 13 | 29
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 13 | 29
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 4 | 11
  White | 4 | 4 | 9 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Score
Description: Average pain score (VAS) 48 hrs postoperatively between the study group and the control. The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. 0 represents no pain, whereas 10 represents unbearable pain.
Time Frame: 48 hours postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | 2mg Dexamethasone | 4mg Dexamethasone
Number analyzed (Participants) | 7 | 9 | 13
units on a scale | 1.49 (0.25) | 1.40 (0.40) | 1.62 (0.35)

2. Secondary Outcome: First Post-Operative Opioid Administration
Description: Time until first dose post-operative opioid administration between the study group and the control
Time Frame: baseline to 48 hrs postoperatively
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Control Group | 2mg Dexamethasone | 4mg Dexamethasone
Number analyzed (Participants) | 7 | 9 | 13
Hours | 22.43 (4.87) | 12.56 (3.58) | 18.25 (4.23)

3. Secondary Outcome: Average Opioid Consumption
Description: Average opioid consumption 48 hrs postoperatively between the study group and the control
Time Frame: from the time of delivery to 48hrs postoperatively
Measure: Mean (Standard Deviation); unit: mg of morphine equivalents
Arm/Group | Control Group | 2mg Dexamethasone | 4mg Dexamethasone
Number analyzed (Participants) | 7 | 9 | 13
mg of morphine equivalents | 37.93 (13.50) | 47.11 (12.44) | 42.38 (9.17)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group | 2mg Dexamethasone | 4mg Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 0/13

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed, due to recruitment challenges related to competing studies in the women and infants center

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT03098420/Prot_SAP_000.pdf